CLINICAL TRIAL: NCT00555984
Title: Effect of Total Intravenous Anesthesia Versus Anesthesia With Volatile Agents on Inflammatory Markers Following Elective Craniotomy for Primary Brain Tumor
Brief Title: Intravenous Anesthesia Versus Anesthesia With Volatile Agents in Elective Craniotomy for Tumors
Acronym: TIVA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision to terminate. No usable data collected
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Case 4306; NCT00524082 (obsolete NCT alias)
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Brain Neoplasms
Keywords: Intracranial tumors; Inflammatory markers; Craniotomy; Postoperative complications
MeSH Terms: conditions — Brain Neoplasms; Postoperative Complications | interventions — Propofol; Remifentanil; Anesthetics, Intravenous; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total Intravenous anesthetic (Active Comparator): Intravenous anesthetics (propofol + remifentanil) for maintenance of General Anesthesia
  Interventions: Drug: Propofol + Remifentanil
- Volatile Anesthetic (Active Comparator): Inhalational anesthetics (sevoflurane+remifentanil) for maintenance of General Anesthesia. Patients receive Sevoflurane as a volatile anesthetic and remifentanil as an IV agent for maintenance of general anesthesia.
  Interventions: Drug: Sevoflurane + Remifentanil

INTERVENTIONS:
Drug: Propofol + Remifentanil — Administered intravenously during surgery for maintenance of General Anesthesia
  Other Names: Intravenous anesthetics
  Arms: Total Intravenous anesthetic
Drug: Sevoflurane + Remifentanil — the (Sevoflurane + Remifentanil) arm: Sevoflurane as inhalational agent and Remifentanil as intravenous agent for maintenance of General Anesthesia
  Other Names: Inhalational anesthetics
  Arms: Volatile Anesthetic

SUMMARY:
If the anesthetic regimen can influence the serum level of inflammatory cytokines and if the levels of cytokines are related to the incidence of post operative complications, these complications may be a function of the anesthetic method. In an effort to find the best anesthetic regimen for patients undergoing craniotomy for intracranial tumors, the researchers will compare the effect of volatile anesthetic with that of total intravenous anesthesia (TIVA) on cytokine levels. The researchers will also compare the composite incidence of some common major post-operative complications after craniotomy for intracranial malignancy.

DETAILED DESCRIPTION:
This is a randomized blinded clinical trial. Patients will be randomized into one of two groups. One group will receive a volatile anesthetic (sevoflurane)while the other group will receive intravenous anesthetics (propofol + remifentanil) for maintenance of General Anesthesia.

The anesthesia team will know the result of randomization at induction. Postoperative data will be gathered by research personnel who will be blinded to the anesthetic method used. Patients will be blinded to the anesthetic they receive until after the 4-week outcomes are collected, when they will have the option to be unblinded.

Peripheral blood samples will be taken a total of 7 times; pre-induction to anesthesia, 15 minutes after surgical positioning, after the tumor is extracted, and at 6,12,18, and 24 hours after emergence from anesthesia.

Patients will be called for follow up every week for 4 weeks following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia for elective surgical excision of a primary brain tumor
* Age: Older than 18
* New and recurrent cases will be included

Exclusion Criteria:

* Patient refusal
* Emergency craniotomy
* Craniotomy after head injuries or intracranial bleeding
* Patients with active inflammatory processes such as infection or immunologic illnesses known to increase baseline immunologic markers
* Preoperative diagnosis of DVT by lower extremity ultrasound or symptoms
* Preoperative pulmonary infiltrative disease (pulmonary fibrosis, sarcoid, etc.)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To study inflammatory changes associated with these two different anesthetic techniques | 24 hours post-operatively

SECONDARY OUTCOMES:
Because of the linkage between cytokines, thrombotic disease, tissue inflammation and brain edema, we plan to monitor a composite outcome derived from occurrence of DVT, PE, new neurologic deficit, postoperative infection and respiratory failure | 4 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Avitsian, MD, Principal Investigator — The Cleveland Clinic; Armin Schubert, MD, MBA, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated early